CLINICAL TRIAL: NCT05060016
Title: A Phase 2 Study Evaluating the Efficacy, Safety, Tolerability, and Pharmacokinetics of Tarlatamab in Subjects With Relapsed/Refractory Small Cell Lung Cancer After Two or More Prior Lines of Treatment (DeLLphi-301).
Brief Title: A Phase 2 Study of Tarlatamab in Patients With Small Cell Lung Cancer (SCLC)
Acronym: DeLLphi-301
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20200491; 2024-511837-37 (Other: EU-CTR)
Expanded Access: NCT06064500 (Approved for marketing)
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Relapsed/Refractory Small Cell Lung Cancer
Keywords: Small Cell Lung Cancer; SCLC; AMG 757; Tarlatamab; IMDELLTRA^TM
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Tarlatamab Low Dose (Experimental): Participants will receive the low dose of Tarlatamab.
  Interventions: Drug: Tarlatamab
- Part 1: Tarlatamab High Dose (Experimental): Participants will receive the high dose of Tarlatamab.
  Interventions: Drug: Tarlatamab
- Part 2: Dose Expansion (Experimental): Participants will receive the selected target dose of Tarlatamab based on findings in Part 1.
  Interventions: Drug: Tarlatamab
- Part 3: Modified Monitoring Substudy (Experimental): Participants will receive the selected target dose of Tarlatamab based on findings in Part 1 with reduced Cycle 1 monitoring requirements.
  Interventions: Drug: Tarlatamab

INTERVENTIONS:
Drug: Tarlatamab — Intravenous (IV) infusion

SUMMARY:
The main aim of this study is to:

* evaluate safety and efficacy (per Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST 1.1] by investigator) of 2 dose levels of tarlatamab for Part 1 only
* evaluate anti-tumor activity of tarlatamab as determined by objective response rate (ORR) per RECIST 1.1 by blinded independent central review (BICR) for Part 1 and 2
* evaluate safety of reduced mandatory monitoring period in Cycle 1 at selected dose of tarlatamab for Part 3

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided informed consent/assent prior to initiation of any study specific activities/procedures.
* Male and female participants ≥ 18 years of age (or legal adult age within country) at the time of signing the informed consent.
* Histologically or cytologically confirmed relapsed/refractory SCLC
* Participants who progressed or recurred following 1 platinum-based regimen and at least 1 other prior line of therapy.
* Participants willing to provide archived tumor tissue samples or willing to undergo pretreatment tumor biopsy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 1.
* Minimum life expectancy of 12 weeks.
* Measurable lesions as defined per RECIST 1.1 within 21 days prior to the first dose of tarlatamab.
* Participants with treated brain metastases are eligible provided they meet defined criteria.

Exclusion Criteria:

Disease Related

* Untreated or symptomatic brain metastases and leptomeningeal disease.
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Participants who experienced recurrent pneumonitis (grade 2 or higher) or severe, life-threatening immune-mediated adverse events or infusion-related reactions including those that lead to permanent discontinuation while on treatment with immuno-oncology agents.
* Unresolved toxicity from prior anti-tumor therapy, defined as per protocol.

Other Medical Conditions

* History of other malignancy within the past 2 years, with exceptions
* Myocardial infarction and/or symptomatic congestive heart failure (New York Heart Association > class II) within 12 months of first dose of tarlatamab.
* History of arterial thrombosis (eg, stroke or transient ischemic attack) within 12 months of first dose of tarlatamab.
* Participant with symptoms and/or clinical signs and/or radiographic signs that indicate an acute and/or uncontrolled active systemic infection within 7 days prior to the first dose of tarlatamab.
* Presence of any indwelling line or drain.
* History of hypophysitis or pituitary dysfunction.
* Exclusion of hepatitis infection based on the results and/or criteria per protocol.
* Major surgery within 28 days of first dose of tarlatamab.
* History or evidence of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection. Subject is eligible if no acute symptoms of coronavirus disease 2019 (COVID-19) within 14 days prior to first dose of tarlatamab (counted from day of positive test for asymptomatic subjects).

Prior/Concomitant Therapy

* Participant received prior therapy with tarlatamab.
* Prior anti-cancer therapy within 28 days prior to first dose of tarlatamab.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of tarlatamab.
* The following vaccines (live and live-attenuated vaccines) are excluded during the following study periods:

  1. Screening and during study treatment: Live and live-attenuated vaccines are prohibited within 28 days prior to the first dose of tarlatamab and for the duration of the study. Live viral non-replicating vaccine (e.g. Jynneos) for Monkeypox infection is allowed during the study (except during cycle 1) in accordance with local standard of care and institutional guidelines.
  2. End of study treatment: Live and live-attenuated vaccines can be used when at least 42 days (5X half-life of tarlatamab) have passed after the last dose of tarlatamab.

Other Exclusions

* Female participants of childbearing potential unwilling to use protocol specified method of contraception during treatment and for an additional 60 days after the last dose of tarlatamab.
* Female participants who are breastfeeding or who plan to breastfeed while on study through 60 days after the last dose of tarlatamab.
* Female participants planning to become pregnant while on study through 60 days after the last dose of tarlatamab.
* Female participants of childbearing potential with a positive pregnancy test assessed at screening and/or day 1 by a highly sensitive urine or serum pregnancy test.
* Male participants with a female partner of childbearing potential who are unwilling to practice sexual abstinence (refrain from heterosexual intercourse) or use contraception during treatment and for an additional 60 days after the last dose of tarlatamab.
* Male participants with a pregnant partner who are unwilling to practice abstinence or use a condom during treatment and for an additional 60 days after the last dose of tarlatamab.
* Male participants unwilling to abstain from donating sperm during treatment and for an additional 60 days after the last dose of tarlatamab.
* Participant has known sensitivity to any of the products or components to be administered during dosing.
* Participant likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures.
* History or evidence of any other clinically significant disorder, condition or disease determined by the investigator or Amgen physician.

Specific Exclusions to Part 3

* Participants unable to remain within one hour of study site for 48 hours after infusion of tarlatamab on Cycle 1 Day 1 and Cycle 1 Day 8.
* Participants unable to remain within one hour of any hospital for 72 hours after infusion of tarlatamab on Cycle 1 Day 1 and Cycle 1 Day 8.
* Unable to identify home companion who will cohabitate with participant for 72 hours after infusion of tarlatamab on Cycle 1 Day 1 and Cycle 1 Day 8.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Part 1 Only: Objective Response (OR) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by Investigator | Up to a maximum of 61 months
Part 1 and Part 3 Only: Number of Participants who Experience One or More Treatment-emergent Adverse Events | Up to a maximum of 61 months
Part 1 Only: Serum Concentrations of Tarlatamab | Up to a maximum of 24 months
Part 1 and Part 2 Only: Objective Response (OR) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by Blinded Independent Central Review (BICR) | Up to a maximum of 61 months

SECONDARY OUTCOMES:
Duration of Response (DOR) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by Blinded Independent Central Review (BICR) | Up to a maximum of 73 months
Disease Control (DC) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by Blinded Independent Central Review (BICR) | Up to a maximum of 73 months
Duration of Disease Control (DC) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by Blinded Independent Central Review (BICR) | Up to a maximum of 73 months
Progression-free Survival (PFS) Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by Blinded Independent Central Review (BICR) | Up to a maximum of 73 months
Objective Response (OR) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by Investigator | Up to a maximum of 73 months
Duration of Response (DOR) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by Investigator | Up to a maximum of 73 months
Disease Control (DC) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by Investigator | Up to a maximum of 73 months
Duration of Disease Control (DC) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by Investigator | Up to a maximum of 73 months
Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by Investigator | Up to a maximum of 73 months
Overall Survival (OS) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by Investigator | Up to a maximum of 73 months
Number of Participants who Experience One or More Treatment-emergent Adverse Events | Up to a maximum of 73 months
Serum Concentrations of Tarlatamab | Up to a maximum of 24 months
Number of Participants who Experience Anti-Tarlatamab Antibody Formation | Up to a maximum of 73 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (80):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Christiana Care Health Services, Newark, Delaware
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - Dana Farber - Harvard Cancer Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Dartmouth Hitchcock Medical Center, Hanover, New Hampshire
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Comprehensive Cancer Research Center, Winston-Salem, North Carolina
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University of Pittsburgh Medical Center Cancer Pavillion, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - West Virginia University Health Sciences Center, Morgantown, West Virginia
- Austria (2):
  - Universitaetsklinikum Krems, Krems
  - Landeskrankenhaus Salzburg, Salzburg
- Belgium (3):
  - Universitair Ziekenhuis Gent, Ghent
  - Grand Hopital de Charleroi - Site Saint Joseph, Gilly
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
- Rigshospitalet, Copenhagen, Denmark
- France (7):
  - Centre Hospitalier Universitaire Nord, Marseille
  - Institut Curie, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Rennes - Hopital Pontchaillou, Rennes
  - Centre Hospitalier Universitaire de Strasbourg - Nouvel Hopital Civil, Strasbourg
  - Centre Hospitalier Universitaire de Toulouse - Hopital Larrey, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (3):
  - Universitaetsklinikum Koeln, Cologne
  - LungenClinic Grosshansdorf GmbH, Großhansdorf
  - Universitaetsklinikum Wuerzburg, Würzburg
- Greece (8):
  - Henry Dunant Hospital Center, Athens
  - Sotiria General Hospital, Athens
  - Metropolitan Hospital, Athens
  - University Hospital of Heraklion, Heraklion - Crete
  - General Hospital of Patras Agios Andreas, Pátrai
  - Theagenion Cancer Hospital, Thessaloniki
  - Euromedica General Clinic of Thessaloniki, Thessaloniki
  - Agios Loukas Clinic, Thessaloniki
- Italy (3):
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Istituti Fisioterapici Ospitalieri Regina Elena San Gallicano, Rome
  - Azienda Socio Sanitaria Territoriale dei Sette Laghi Ospedale di Circolo e Fondazione Macchi, Varese
- Japan (7):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Okayama University Hospital, Okayama, Okayama-ken
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-ku, Tokyo
  - Wakayama Medical University Hospital, Wakayama, Wakayama
- Netherlands (2):
  - Leids Universitair Medisch Centrum, Leiden
  - Erasmus Medisch Centrum, Rotterdam
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Centra Medyczne Medyceusz Sp zoo, Lodz
  - Mazowieckie centrum leczenia, Otwock
- Portugal (5):
  - Hospital da Luz, SA, Lisbon
  - Hospital CUF Descobertas, Lisbon
  - Centro Hospitalar Universitario do Porto EPE - Hospital de Santo Antonio, Porto
  - Hospital Cuf porto, Porto
  - Instituto Portugues de Oncologia do Porto Francisco Gentil, EPE, Porto
- National Cancer Centre Singapore, Singapore, Singapore
- South Korea (6):
  - National Cancer Center, Goyang-si Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Yonsei University Health System Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung medical center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
- Spain (8):
  - Hospital Regional Universitario de Malaga, Málaga, Andalusia
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Instituto Catalan de Oncologia Hospital Duran i Reynals, L'Hospitalet de Llobregat, Catalonia
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia, Valencia
  - Hospital Universitario 12 de Octubre, Madrid
- Hopitaux Universitaires de Geneve, Geneva, Switzerland
- Taiwan (2):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (2):
  - Sarah Cannon Research Institute UK, London
  - Christie Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Ahn MJ, Cho BC, Felip E, Korantzis I, Ohashi K, Majem M, Juan-Vidal O, Handzhiev S, Izumi H, Lee JS, Dziadziuszko R, Wolf J, Blackhall F, Reck M, Bustamante Alvarez J, Hummel HD, Dingemans AC, Sands J, Akamatsu H, Owonikoko TK, Ramalingam SS, Borghaei H, Johnson ML, Huang S, Mukherjee S, Minocha M, Jiang T, Martinez P, Anderson ES, Paz-Ares L; DeLLphi-301 Investigators. Tarlatamab for Patients with Previously Treated Small-Cell Lung Cancer. N Engl J Med. 2023 Nov 30;389(22):2063-2075. doi: 10.1056/NEJMoa2307980. Epub 2023 Oct 20. PMID 37861218
- [Background] Ahn MJ, Cho BC, Felip E, Korantzis I, Ohashi K, Majem M, Juan-Vidal O, Handzhiev S, Izumi H, Lee JS, Dziadziuszko R, Wolf J, Blackhall F, Reck M, Alvarez JB, Hummel HD, Dingemans AC, Sands J, Akamatsu H, Owonikoko TK, Ramalingam SS, Borghaei H, Johnson ML, Huang S, Mukherjee S, Minocha M, Jiang T, Martinez P, Anderson ES, Paz-Ares L. Plain language summary: tarlatamab for patients with previously treated small cell lung cancer. Future Oncol. 2024 Dec;20(40):3355-3364. doi: 10.1080/14796694.2024.2402152. Epub 2024 Nov 12. PMID 39530627
- [Background] Hummel HD, Ahn MJ, Blackhall F, Reck M, Akamatsu H, Ramalingam SS, Borghaei H, Johnson M, Dirnberger F, Cocks K, Huang S, Mukherjee S, Paz-Ares L. Patient-Reported Outcomes for Patients with Previously Treated Small Cell Lung Cancer Receiving Tarlatamab: Results from the DeLLphi-301 Phase 2 Trial. Adv Ther. 2025 Apr;42(4):1950-1964. doi: 10.1007/s12325-025-03136-4. Epub 2025 Mar 3. PMID 40025391
- [Background] Kong S, Minocha M, Chen PW, Martinez P, Anderson ES, Parkes A, Houk BE, Lin CW. Population Pharmacokinetics of Tarlatamab, a Half-Life Extended DLL3-Directed Bispecific T-Cell Engager in Patients with Previously Treated Small Cell Lung Cancer. Clin Pharmacokinet. 2025 May;64(5):729-741. doi: 10.1007/s40262-025-01499-z. Epub 2025 Apr 22. PMID 40261494
- [Background] Ahn MJ, Cho BC, Ohashi K, Izumi H, Lee JS, Han JY, Chiang CL, Huang S, Hamidi A, Mukherjee S, Xu KL, Akamatsu H. Asian Subgroup Analysis of Patients in the Phase 2 DeLLphi-301 Study of Tarlatamab for Previously Treated Small Cell Lung Cancer. Oncol Ther. 2025 Dec;13(4):1041-1054. doi: 10.1007/s40487-025-00372-0. Epub 2025 Sep 4. PMID 40908346
- [Background] Chen PW, Minocha M, Kong S, Jiang T, Anderson ES, Parkes A, Martinez P, Houk BE, Lin CW. Tarlatamab Exposure-Efficacy and Exposure-Safety Relationships to Inform Dose Selection in Patients with Small Cell Lung Cancer. Clin Cancer Res. 2025 Nov 14;31(22):4688-4697. doi: 10.1158/1078-0432.CCR-25-2134. PMID 40928991
- [Background] Dirnberger F, Wang J, King-Kallimanis B, Cocks K, Skingley G, Clarke N, Huang S, Mukherjee S, Koller M. Derivation of Meaningful Change Thresholds for European Organization for Research and Treatment of Cancer QLQ-C30 and QLQ-LC13 in Patients With Small-Cell Lung Cancer. Value Health. 2026 Feb;29(2):223-232. doi: 10.1016/j.jval.2025.09.011. Epub 2025 Sep 25. PMID 41015335
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com